CLINICAL TRIAL: NCT00633061
Title: Phase II Study on the Identification and Treatment of Clinically Silent Catheter-Related Deep Vein Thrombosis in Children With Cancer
Brief Title: Identification and Treatment of Clinically Silent Catheter-Related Deep Vein Thrombosis in Children With Cancer
Acronym: DVT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Futility; unable to complete screening due to clinical practice change
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23HL084097 (NIH); STU12207-062 (Other: University of Texas-Southwestern Medical Center)
Record Dates: First submitted 2008-02-24; First posted 2008-03-11 (Estimated); Results first posted 2019-03-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Childhood Cancer; Central Venous Catheters; Deep Vein Thrombosis; Catheter-related Infection; Catheter-related Occlusion
Keywords: Childhood Cancer; Central Venous Catheter; Deep Vein Thrombosis; Catheter-related Infection; Catheter-related Occlusion
MeSH Terms: conditions — Neoplasms; Venous Thrombosis; Catheter-Related Infections | interventions — Enoxaparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A-randomized to treatment (Experimental): Patients diagnosed with asymptomatic catheter-related DVT who are randomized to treatment with enoxaparin for 6 weeks
  Interventions: Drug: Enoxaparin
- B-randomized to close (No Intervention): Patients diagnosed with asymptomatic catheter-related DVT who are randomized to close observation for 6 weeks

INTERVENTIONS:
Drug: Enoxaparin — Lovenox ® is a sterile aqueous solution containing enoxaparin sodium, a low molecular weight heparin. It is given as a subcutaneous injection twice daily. Dose of enoxaparin (Lovenox ®) will be 1 mg/kg every 12 hours for children >2 months and 1.5 mg/kg every 12 hours for infants <2 months. Duration of treatment is 6 weeks.
  Other Names: Lovenox
  Arms: A-randomized to treatment

SUMMARY:
The primary hypothesis of this study is that occult catheter-related DVT in children with cancer is common and directly contributes to development of serious catheter complications, specifically bacteremia/fungemia and/or recurrent occlusion of the catheter tip. Accordingly, anticoagulant treatment of clinically silent (occult) DVT will reduce rates of catheter-related infection and occlusion, delays in therapy and need for catheter replacement.

DETAILED DESCRIPTION:
This is a two-part study with an initial diagnosis component followed by a treatment component. The number of subjects to be consented for the diagnosis component is 350, and 50 for the treatment portion (25 on the observation arm, and 25 for enoxaparin treatment).

Study Procedures:

Patients diagnosed with cancer at the Center for Cancer and Blood Disorders will have a catheter inserted for cancer related treatment. After insertion, eligible patients who provide consent will be enrolled in the diagnosis component of the study. The principal investigator and research team will monitor for catheter complications (occlusion and bacteremia/fungemia). After two complications, participants will be screened for occult central venous catheter (CVC)-related DVT by contrast venography, ultrasonography, or magnetic resonance venography. If DVT is not diagnosed, participant will go off the study. If DVT is diagnosed, participant will be asked to consent to enroll in the treatment study. After enrollment, participant is randomized between the two arms of observation and enoxaparin treatment. After 6 weeks, patients will have another image; this represents the end of treatment period. After the follow-up imaging, patients will be monitored for 10 weeks to obtain primary outcomes. Once a primary outcome (progression to symptomatic DVT or pulmonary embolism (PE), blood stream infection or catheter removal) is achieved the participants can be treated with anticoagulation again if necessary, but primary oncologist will determine treatment.

Analysis:

The hypothesis is that the enoxaparin treatment group will have a median adverse catheter event free survival time of 12 weeks versus 4 weeks for the control group with a hazard ration of 0.4. A total sample size of 50 (25 in each arm) will detect such a difference with 90% power at an α=0.05. If there is a drop out rate of 10% in each arm, a difference can still be detected with 80% power.

Approximately 200 to 250 patients are diagnosed with cancer each year at Children's Medical Center Dallas, and based on prior institutional experience, two-thirds will have catheters inserted to facilitate chemotherapy. However, one-quarter of these patients have brain tumors and are not eligible due to the potential increased risk of intracranial hemorrhage with anticoagulation. There will be 100 patients each year who are at risk for CVC-related DVT. Based on previous studies, up to 50% of patients should develop occult DVT; however, only 35% of patients will likely be screened with radiographic imaging. Approximately 17 patients a year enrolled in the diagnosis study may be diagnosed with DVT and eligible for randomization. Therefore, total enrollment will be completed in approximately 3 years with an additional 4 months necessary to complete the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of cancer
2. Age ≤ 18 years
3. First tunneled central venous catheter (implanted port or external) inserted in the upper venous system (subclavian, brachiocephalic, or jugular vein) within the previous 2 weeks
4. Catheter expected to be in place for duration of chemotherapy (≥ 3 months)
5. History of no more than one catheter complication (occlusion or infection)

Exclusion Criteria:

1. Prior history of DVT
2. Currently receiving an anticoagulant or anti-platelet agents on a daily basis
3. Diagnosis of high grade malignant brain tumor or metastasis to the brain
4. Clinical signs/symptoms of DVT
5. Clinical signs/symptoms of Pulmonary embolism
6. Renal failure
7. Recent major hemorrhage

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 136 (Actual)
Dates: Start 2008-06 (Actual); Primary Completion 2011-06 (Actual); Study Completion 2011-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janna Journeycake, MD, Principal Investigator — University of Texas
Locations (1):
- Children's Medical Center, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from June 2008 to December 2010. For arm A, we screened 486 children and enrolled 136. 68 patients were eligible and not enrolled and 282 were ineligible.
  No patient was eligible for Arm B of this study
Groups:
- A-Prosepctive Screening for Asymptomatic DVT: Patients </=18 years of age with cancer and a first indwelling catheter expected to be in place for 3 months are enrolled. They are screened with either contrast venogram or ultrasound for asymptomatic catheter-related DVT if they have had at least 2 complications including line occlusion requiring tpa or catheter infection that did not result in removal of the line. If they have a positive screening study they are eligible for Arm B
- B-Randomized Clinical Trail for Treatment: Patients diagnosed with asymptomatic catheter-related DVT who are randomized to between enoxaparin or close observation for 6 weeks
Period: Overall Study
Arm/Group | A-Prosepctive Screening for Asymptomatic DVT | B-Randomized Clinical Trail for Treatment
Started | 136 (Study was on hold for 2 months for continuing review) | 0
Met Criteria for Imaging | 25 | 0
Had Prior Thrombosis Identified | 25 | 0
Completed | 50 | 0
Not Completed | 86 | 0
Not completed — Study closed | 86 | 0

BASELINE CHARACTERISTICS:
Population: No patient from arm A was eligible to enroll in Arm B.
Groups:
- A-Prosepctive Screeing for Asymptomatic DVT: Patients diagnosed with asymptomatic catheter-related DVT who are randomized to treatment with enoxaparin for 6 weeks
  Enoxaparin: Lovenox ® is a sterile aqueous solution containing enoxaparin sodium, a low molecular weight heparin. It is given as a subcutaneous injection twice daily. Dose of enoxaparin (Lovenox ®) will be 1 mg/kg every 12 hours for children >2 months and 1.5 mg/kg every 12 hours for infants <2 months. Duration of treatment is 6 weeks.
- B-Randomized Clinical Trail for Treatment: Patients diagnosed with asymptomatic catheter-related DVT who are randomized to close observation for 6 weeks
- Total: Total of all reporting groups
Arm/Group | A-Prosepctive Screeing for Asymptomatic DVT | B-Randomized Clinical Trail for Treatment | Total
Number analyzed (Participants) | 136 | 0 | 136
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 136 |  | 136
  Between 18 and 65 years | 0 |  | 0
  >=65 years | 0 |  | 0
Age, Continuous [Mean (Full Range); unit: years] | 10 [1 to 18] |  | 10 [1 to 18]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69 |  | 69
  Male | 67 |  | 67
Region of Enrollment [Number; unit: participants]
  United States | 136 |  | 136

OUTCOME MEASURES:

1. Primary Outcome: Composite Endpoint for Arm B of the Study: Catheter Removal, Signs and Symptoms of DVT or PE, OR Bacteremia/Fungemia
Description: catheter removal, signs and symptoms of DVT or PE, OR bacteremia/fungemia
Time Frame: 16 weeks
Population: No patient was enrolled on the randomized clinical trial (arm B) after being on the prospective screening trial (Arm A)
Groups:
- B-Randomized Clinical Trail for Treatment: Patients diagnosed with asymptomatic catheter-related DVT who are randomized to close observation or treatment with enoxaparin
Arm/Group | A- Prospective Screening for Asymptomatic Catheter-related DVT | B-Randomized Clinical Trail for Treatment
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Bleeding Complications Associated With Enoxaparin Therapy, Need for Additional Platelets
Description: Bleeding complications associated with enoxaparin therapy, need for additional platelets
Time Frame: 6 weeks
Population: Since no patient was enrolled on Arm B of this study, there is no analysis of bleeding.
Groups:
- A: Prospectvie Screening for Asymptomatic Catheter-related DVT: Patients </=18 years of age with cancer and a first indwelling catheter expected to be in place for 3 months are enrolled. They are screened with either contrast venogram or ultrasound for asymptomatic catheter-related DVT if they have had at least 2 complications including line occlusion requiring thrombolysis or catheter infection that did not result in removal of the line. If they have a positive screening study they are eligible for Arm B
- B-randomized Treatment Trail: Patients diagnosed with asymptomatic catheter-related DVT who are randomized to close observation or enoxaparin to treat asymptomatic DVT
Arm/Group | A: Prospectvie Screening for Asymptomatic Catheter-related DVT | B-randomized Treatment Trail
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Groups:
- A-Prospective Screening for Asymptomatic Catheter-related DVT: Patients </=18 years of age with cancer and a first indwelling catheter expected to be in place for 3 months are enrolled. They are screened with either contrast venogram or ultrasound for asymptomatic catheter-related DVT if they have had at least 2 complications including line occlusion requiring thrombolysis or catheter infection that did not result in removal of the line. If they have a positive screening study they are eligible for Arm B
- B-Randomized Clinical Trial: Patients diagnosed with asymptomatic catheter-related DVT who are randomized to close observation vs enoxaparin for 6 weeks
Arm/Group | A-Prospective Screening for Asymptomatic Catheter-related DVT | B-Randomized Clinical Trial
All-Cause Mortality (participants affected / at risk) | 0/136 | 0/0
Serious Adverse Events (participants affected / at risk) | 16/136 | 0/0
Other Adverse Events (participants affected / at risk) | 0/136 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A-Prospective Screening for Asymptomatic Catheter-related DVT (N=136) | B-Randomized Clinical Trial (N=0)
Thrombosis (Vascular disorders) | 7 (7) | 0 — Any thrombotic event
removal of indwelling catheter for reasons other than end of therapy (Vascular disorders) | 9 (9) | 0

LIMITATIONS AND CAVEATS:
Study terminated early for lack of accrual on Arm B (randomized trial). No patient enrolled on Arm A (screening study) were eligible. Standard treatment of asymptomatic catheter-related DVT changed in 2010, favoring treatment with enoxaparin.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No